CLINICAL TRIAL: NCT04405973
Title: Clinical Scores for Outcome Prediction in Patients With Severe COVID-19 Pneumonia Requiring Extracorporeal Membrane Oxygenation - a Retrospective Multi-center Registry Study
Brief Title: Clinical Scores for Outcome Prediction in Patients With Severe COVID-19 Pneumonia Requiring ECMO
Status: Completed | Type: Observational
Sponsor: Dr. Alexander Supady (Other)
Responsible Party: Sponsor-Investigator, Dr. Alexander Supady, Attending Physician - Oberarzt, University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Other Study IDs: EK-FR 329/20
Record Dates: First submitted 2020-05-25; First posted 2020-05-28 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: COVID-19; SARS-CoV 2; Extracorporeal Membrane Oxygenation; ARDS
Keywords: ECMO; ARDS; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 ARDS, vv-ECMO: All patients in the study centers with diagnosed COVID-19 infection (PCR proven) and treatment with vv-ECMO
  Interventions: Device: vv-ECMO

INTERVENTIONS:
Device: vv-ECMO — vv-ECMO required in severe COVID-19 ARDS

SUMMARY:
The prognosis of patients with severe COVID-19 disease, whose lungs are so severely diseased that they need to be supported by veno-venous ECMO (extracorporeal membrane oxygenation), is difficult to assess so far. Previously published data from studies, case reports and case series describe a very high mortality in this patient collective. The significance of established clinical prognostic cores in this patient population has not been systematically investigated. This is aggravated by the fact that even at very specialized centers only very few patients from this collective are (can be) treated, so that valid investigations are only possible in a multicenter patient collective. In this registry study, all patients diagnosed with COVID-19 and treated with vv-ECMO in the centers participating in the study should be retrospectively examined. The primary aim of the study is to investigate 30-day survival, secondary objectives include the analysis of different clinical scores at the time of ECMO implantation.

DETAILED DESCRIPTION:
In December 2019, a series of unexplained cases of pneumonia in the city of Wuhan in China has come to light. In virologic analyses of samples from the patients' deep respiratory tract, a novel coronavirus was isolated (first named 2019-nCoV, then SARS-CoV-2). The disease spread rapidly in the city of Wuhan in early 2020 and soon beyond. On 30 January 2020, the Director-General of the World Health Organization (WHO) declared the outbreak a public health emergency of international concern, and on 11 March 2020, the World Health Organization declared the virus a pandemic.

In humans, an infection with the virus can cause respiratory tract infections or even very severe pneumonia - these often end fatally, especially in old and pre-diseased patients. Due to the novelty of the virus, the data basis for therapy is very limited. To date, there are no clinical data for an effective specific therapy, nor is there a vaccination against the virus available, so that therapy, especially intensive care treatment for very severe courses, must concentrate only on supportive treatment of lung failure and other complications.

The virus is highly contagious and infection results in a relevant number of deaths. Due to very uncertain data on the spread of the virus in the population, it is difficult to estimate the mortality rate - the case fatality rate is about 4% based on the known case numbers.

In reports on the treatment of the first cases in Wuhan (Hubei Province, China) in January 2020, the need for intensive care treatment is described for about a quarter of the inpatient cases, 10-17% had to be ventilated invasively, and veno-venous extracorporeal membrane oxygenation (vv-ECMO) was necessary in 2-4% of the inpatient cases. Patients requiring ECMO have a high mortality rate in the studies published, so far. Recommendations for initiation of ECMO in COVID-19 are being developed, though under continuous review.

Currently, little is known to guide clinicians in the choice of patients eligible for ECMO in COVID-19, nor about the best time point for initiation of ECMO or the value of established clinical scores for the prediction of the outcome of patients.

The aim of the study is to investigate survival in COVID-19 patients requiring vv-ECMO support. Furthermore, the accuracy of clinical scores, established in intensive care medicine for the prediction of outcome in severely ill patients will be assessed. Finally, time to extubation from ventilation and time to ECMO-explantation will be evaluated. The study design is a single-arm retrospective multi-center registry; therefore, no comparator will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patient admitted to ICU
* initiation of vv-ECMO
* definite SARS-CoV-2-infection

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All COVID-19-patients treated on an ICU at the participating centers and requeiring vv-ECMo support
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
overall survival | 30 days
  time from ECMO-implantation to death

SECONDARY OUTCOMES:
duration of ECMO treatment | 30 days
  time from ECMO-implantation to ECMO-explantation
duration of ventilation treatment | 30 days
  time from ECMO-implantation to extubation
duration of initiation of ECMO treatment to ICU discharge | 30 days
  time from ECMO-implantation to ICU-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Supady, MD, MPH, Principal Investigator — University Clinic Freiburg
Locations (1):
- University Clinic Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No